CLINICAL TRIAL: NCT05674916
Title: Effect of a Point-Of-Care Ultrasound-Driven vs Standard Diagnostic Pathway on 24-Hour Hospital Stay in Emergency Department Patients With Dyspnea - a Randomized Controlled Trial
Brief Title: Point-Of-Care Ultrasound-Driven vs Standard Diagnostic Pathway in Emergency Department Patients With Dyspnea
Acronym: POCUS PATHWAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Stig Holm Ovesen, MD, Principal Investigator, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: pocuspathway
Record Dates: First submitted 2022-12-16; First posted 2023-01-09 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Dyspnea
Keywords: Point-of-care Ultrasound; Emergency Medicine; Diagnostic pathways
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Point-of-care ultrasound-driven diagnostic pathway (Experimental): The intervention is focused lung and cardiac ultrasound performed as an extension to physical examinations plus diagnostic decision recommendations based on those test results (a point-of-care ultrasound-driven diagnostic pathway). Final decision on next-line imaging and further diagnostic testing should incorporate history and other physical examinations and will remain upon the treating physicians' discretion.
  Interventions: Diagnostic Test: Point-of-care ultrasound-driven diagnostic pathway
- Standard diagnostic pathway (No Intervention): Standard diagnostic pathway will include, but not be limited to, blood samples, blood gases, electrocardiogram, and chest x-ray. Focused lung and cardiac ultrasound cannot be performed while the patients stay in the emergency department.

INTERVENTIONS:
Diagnostic Test: Point-of-care ultrasound-driven diagnostic pathway — Focused lung ultrasound will include 8 zones (anterior and lateral) and evaluate pneumothorax, interstitial syndrome, lung consolidation, and pleural effusion. Focused cardiac ultrasound will include four views (subxiphoid four-chamber view, parasternal long-axis view, parasternal short-axis view, and apical four-chamber view) and evaluate pericardial fluid, right ventricle dilation, and left ventricular systolic contractility.
  Arms: Point-of-care ultrasound-driven diagnostic pathway

SUMMARY:
The POCUS PATHWAY-trial is a multi-center, randomized, investigator-initiated, open labelled, pragmatic, controlled trial of a point-of-care ultrasound-driven diagnostic pathway vs standard diagnostic pathway in dyspneic emergency department patients. The primary outcome will be 24-hour hospital stay and 642 patients will be included. Key secondary outcomes include overall hospital length of stay, image resources, and 72-hour revisits.

ELIGIBILITY:
Inclusion Criteria:

1. Emergency department contact
2. Age ≥ 18 years
3. Chief complaint is Dyspnea
4. Including physician present

Exclusion Criteria:

1. Fulfilling of criteria for coded rapid-response teams (i.e., trauma, surgical or medical emergencies).
2. Prior focused lung or focused cardiac ultrasound in the current emergency department stay
3. Prior enrollment in the trial
4. Unable to consent
5. Non Danish-speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
24-hour hospital stay | From date of hospital admission until the date of first documented hospital discharge, assessed up to 24 hours.
  Proportion of patients with a hospital lenght-of-stay of less than 24 hours.

SECONDARY OUTCOMES:
Hospital length-of-stay | From date of hospital admission until the date of first documented hospital discharge, assessed up to 3 months.
  Hospital length-of-stay will secondarily be analyzed using time-to-event analysis.
Image resources | From date of hospital admission until the date of first documented hospital discharge, assessed up to 3 months.
  Image resources will be presented as a composite absolute number and incidence proportion counting the cumulative number of participants having received any of the following imaging techniques during the current hospital stay: chest x-rays, echocardiography, computed tomography (CT) angiography, and CT thorax.
Number of participants with the composite outcome of 72-hour revisits and overall mortality | From date of hospital admission until 72 hours after the date of first documented hospital discharge, assessed up to 3 months.
  72-hour revisits will be defined as a composite outcome including any unplanned hospital stay within 72 hours from the previous hospital discharge, in-hospital mortality, and mortality within 72 hours from the previous hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Stig H Ovesen, Principal Investigator — Aarhus University Hospital
Locations (9):
- Denmark (9):
  - Herlev Hospital, Herlev, Capital Denmark Region
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Gødstrup Regional Hospital, Gødstrup, Central Jutland
  - Horsens Regional Hospital, Horsens, Central Jutland
  - Viborg Regional Hospital, Viborg, Central Jutland
  - University Hospital of Southern Denmark, Esbjerg, Esbjerg, Region Syddanmark
  - Odense University Hospital, Odense, Region Syddanmark
  - Zealand University Hospital, Køge, Køge, Zealand Denmark Region
  - Slagelse Hospital, Slagelse, Zealand Denmark Region

IPD SHARING:
Plan to Share IPD: Yes
Six months after the publication of the last results, all de-identified individual patient data will be made available for data sharing.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: There will be no predetermined end date for the data sharing.
Access Criteria: Data will be available for any research purpose to all interested parties who have approval from an independent review committee and who have a methodological sound proposal as determined by the steering committee of the current trial. Only the methodological qualities and not the purpose or objective of the proposal will be considered. Interested parties will be able to request the data by contacting the principal investigator.

REFERENCES:
- See also: Trial website — https://pocuspathway.org/